CLINICAL TRIAL: NCT03499613
Title: Spinal Kinematics in Chronic Low Back Pain: a Cohort Study
Brief Title: Spinal Kinematics in Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: University of Lausanne Hospitals (Other); University of Lausanne (Other)
Responsible Party: Sponsor
Other Study IDs: LBPKINCOH2017
Record Dates: First submitted 2018-03-14; First posted 2018-04-17 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Chronic Low Back Pain
Keywords: Movement analysis; Spinal kinematics; Muscle activity; Pain-related fear; Rehabilitation; Spine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic low back pain: Patients with chronic low back pain participating to a 3 weeks Multidisciplinary rehabilitation program
  Interventions: Other: Multidisciplinary rehabilitation program

INTERVENTIONS:
Other: Multidisciplinary rehabilitation program — The multimodal rehabilitation program (MRP) based at the University Hospital is an intensive 3-weeks multidisciplinary rehabilitation program. Patients come daily for individual and group treatments, with a total of 100 hours of intervention during 3 weeks. The MRP includes physiotherapy treatments, aiming at improving cardio-vascular endurance, long-term physical activity adherence, proprioception, mobility and strength. Additionally, occupational therapy is mainly focussed on reassuring patients that spinal movements are safe. Finally, psychologists are involved in the MRP to discuss the meaning of LBP, the psychological implications and the patient's resources.

SUMMARY:
Chronic low back pain (CLBP) is one of the most frequent causes for limitations in daily, leisure and work-related activities. Although alterations in spinal motor behavior were consistently reported in CLBP patients, it remains unclear how improvements in spinal motor behavior through rehabilitation treatment affect pain and disability. Psychological factors, such as pain-related fear, were suggested as a possible main cause of spinal motor behavior in CLBP and better understanding their relationships with kinematic and muscle activity alterations is required to enhance care, particularly physiotherapy. Therefore, this study will test CLBP patients before and after a 3 week rehabilitation program to test the hypotheses that: 1) improvements in spinal motor behavior (kinematics and trunk muscle activity) are associated with decreased pain and disability; 2) decrease in pain-related fear is associated with spinal motor behavior improvements.

DETAILED DESCRIPTION:
The research project is a prospective observational cohort study. CLBP patients participating to a 3 weeks' multimodal rehabilitation program will be tested in the motion analysis laboratory before (T1) and after (T2) the program. This program is an intensive 3-weeks multidisciplinary rehabilitation program. Patients come daily for individual and group treatments, with a total of 100 hours of intervention during 3 weeks. The program includes physiotherapy treatments, occupational therapy, psychologists encounters and education session. The programs encompasses a multidimensional view of chronic low back pain. Therefore, this setting is a unique opportunity to improve our understanding of the role of motor behavior alterations in CLBP because it will allow connecting changes in spinal kinematics and muscle activity with changes in pain, disability and pain-related fear.

This project has two aims in relation to motor behavior in patients with CLBP:

The first aim is to analyse the relationship between changes in spinal kinematics and changes in pain and disability during and after a multimodal rehabilitation program. First, changes in spinal kinematics and muscle activity between T1 and T2 will be calculated. The relationship between these changes and changes in pain and disability during the program will be tested. Pain and disability will be also measured at 3 months (T3) and one year (T4) after the program, which will allow to further analyze the relationship between spinal motor behavior and pain and disability.

The second aim concerns the role of pain-related fear, and its decrease, in spinal motor behavior alterations. Consequently, the second aim is to analyse if changes in pain-related fear are associated with changes in spinal kinematics during a multimodal rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* non-specific low back pain (pain from lower ribs to gluteal folds) for more than 3 months
* sufficient French level to understand the instructions for the tests, the information sheet, the consent form and the questionnaires
* both male and female adults will be included
* age more than 18 years old.

Exclusion Criteria:

* pregnancy
* skin allergy to tape
* body mass index (BMI) above 32
* any sign of specific low back pain such as the presence of infection, rheumatologic or neurological diseases, spinal fractures, any known important spinal deformities, previous back surgery that limits spinal mobility, tumours
* high level of pain at the time of experiment that prevents repeated movements (severity and irritability)
* other concomitant pain or condition that could compromise the evaluation of spinal kinematics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain for more than three months participating to a 3 weeks' multidisciplinary rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Spinal kinematics | Change between baseline and week 4
  Range of movement and angular velocity at the lower lumbar, upper lumbar, lower thoracic and upper thoracic joints
Trunk muscle activity | Change between baseline and week 4
  Surface electromyography of paraspinal and abdominal muscles
Pain intensity | Change between baseline and week 4
  Pain intensity will be quantified by the 11-point Numeric Pain Rating Scale. The scale range from 0 (no pain at all) to 10 (worst pain).
Disability | Change between baseline and week 4
  Disability will be quantified by the Patient Specific Functional Scale. The scale assessed three relevant activities for the patient and scores each activity between 0 (impossible to realize the activity) to 10 (capable of doing the activity normally).
Kinesiophobia | Change between baseline and week 4
  Tampa Scale of Kinesiophobia. The total score is between 17 (no kinesiophobia) to 68 (high level of kinesiophobia).
Pain-related fear | Change between baseline and week 4
  Photograph Series of Daily Activities. The score is from 0 (no pain-related fear) to 100 (high levels of pain related fear)
Fear | Change between baseline and week 4
  Fear scale measured before each movement or activity. Score between 0 (no fear) and 10 (high levels of fear).
Pain expectation | Change between baseline and week 4
  Pain expectation scale before each movement or activity. Score between 0 (no pain expected) and 10 (high levels of pain expected).

SECONDARY OUTCOMES:
Disability (ODI) | Baseline (Day 0), week 4, Month 3, Month 12
  Oswestry Disability Questionnaire. Score between 0 (no disability) and 100.
Disability | Month 3, Month 12
  Disability will be quantified by the Patient Specific Functional Scale. The scale assessed three relevant activities for the patient and scores each activity between 0 (impossible to realize the activity) to 10 (capable of doing the activity normally).
Pain intensity | Month 3, Month 12
  Pain intensity will be quantified by the 11-point Numeric Pain Rating Scale. The scale range from 0 (no pain at all) to 10 (worst pain).
Catastrophizing | Baseline (Day 0), week 4, Month 3, Month 12
  Pain Catastrophizing Scale. Score between 0 and 52 (high levels of catastrophizing).
Back Pain Attitudes | Baseline (Day 0), week 4, Month 3, Month 12
  Back Pain Attitudes Questionnaires. Score between 34 (positive attitudes and beliefs) and 170 (negative attitudes and beliefs)
Kinesiophobia | Month 3, Month 12
  Tampa Scale of Kinesiophobia. The total score is between 17 (no kinesiophobia) to 68 (high level of kinesiophobia).
Level of Bothersomeness | Baseline (Day 0), week 4, Month 3, Month 12
  Bothersomeness mesaured with a scale with one question scored from 0 to 4 (Dunn et al, Spine, 2005).
Level of Worry about back pain | Baseline (Day 0), week 4, Month 3, Month 12
  Worry numeric scale. Worry about current back pain is scored from 0 (no worry) to 10 (extremely worried).
Work ability | Baseline (Day 0), Month 3, Month 12
  Work ability. Is back pain limiting the ability to work normally (answer: Yes or No)?
Patient Global Impression of Change | Month 3, Month 12
  This measure is a single-item rating by participants of their improvement with treatment on a 7-point scale that ranges from 'very much improved' (3 points) to 'very much worse' (-3 points) with 'no change' as the mid-point (0 points). The patient will answer this question: "With respect to your low back pain how would you describe yourself now, compared to before the start of the rehabilitation program you did at the University Hospital?"

OTHER OUTCOMES:
Fear of moving | Baseline (Day 0)
  Is there any movement or activity that you don't do or do differently because they are harmful or dangerous for your back ?
Localization of pain | Baseline (Day 0)
  Body chart with localization of pain
Aggravating factors | Baseline (Day 0)
  Which movements or activity increase pain ?
Medication | Baseline (Day 0), week 4, Month 3, Month 12
  Number of medication for low back pain

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lausanne Hospitals, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Christe G, Redhead L, Legrand T, Jolles BM, Favre J. Multi-segment analysis of spinal kinematics during sit-to-stand in patients with chronic low back pain. J Biomech. 2016 Jul 5;49(10):2060-2067. doi: 10.1016/j.jbiomech.2016.05.015. Epub 2016 May 20. PMID 27262182
- [Background] Christe G, Kade F, Jolles BM, Favre J. Chronic low back pain patients walk with locally altered spinal kinematics. J Biomech. 2017 Jul 26;60:211-218. doi: 10.1016/j.jbiomech.2017.06.042. Epub 2017 Jul 5. PMID 28716466